CLINICAL TRIAL: NCT00486707
Title: Questionnaire for Ovarian Cancer Patients Regarding Acceptance and Willingness to Undergo Genetic Testing
Brief Title: Ovarian Cancer Patient Questionnaire on Genetic Testing
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0996
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Questionnaire; Genetic Testing; Survey
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with ovarian cancer
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A questionnaire will be completed.
  Other Names: Survey

SUMMARY:
The objective of this study is to evaluate the willingness of patients with ovarian cancer to undergo genetic testing, given the cost, their understanding and acceptance of genetic testing and the possibility of targeted therapy.

DETAILED DESCRIPTION:
All eligible patients being seen in the Gynecology Center at the M.D. Anderson Cancer Center and at Gynecologic Oncology of Houston for follow-up or a new diagnosis of ovarian cancer will be asked to participate in this study by completing a questionnaire.

This study will end when 400 completed questionnaires have been collected. We estimate that 40-60 ovarian cancer patients are seen in the Gynecology Center at the M.D. Anderson Cancer Center each week and that 20- 40 ovarian cancer patients are seen at Gynecologic Oncology of Houston each week. The completion of 400 questionnaires will provide adequate data to address our question in an expeditious time frame. The initial phase of this study is exploratory and does not involve a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the diagnosis of ovarian cancer.
* Patients must be at least 18 years of age at the time of enrollment.
* Patients must be able to read and write in the English language.

Exclusion Criteria:

* Patients that are unable to speak or write in the English language. Currently, the investigators' resources in genetic counseling are limited. In the future, they plan to expand the questionnaire and study to include additional languages.
* Patients having previously undergone BRCA genetic testing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with a diagnosis of ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Participants' Response to Survey Questions (Yes/No) | 15-20 minutes to complete survey

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Lacour RA, Daniels MS, Westin SN, Meyer LA, Burke CC, Burns KA, Kurian S, Webb NF, Pustilnik TB, Lu KH. What women with ovarian cancer think and know about genetic testing. Gynecol Oncol. 2008 Oct;111(1):132-6. doi: 10.1016/j.ygyno.2008.06.016. Epub 2008 Aug 6. PMID 18684498
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org